CLINICAL TRIAL: NCT04425824
Title: Toripalimab Combine With Rituximab for Treatment of Relapsed Refractory CD20 Positive Diffuse Large B-cell Lymphoma: An Exploratory Small Sample, Phase II, Single-center Clinical Trail
Brief Title: Toripalimab Combine With Rituximab for Treatment of Relapsed Refractory CD20 Positive Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2244
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Diffuse Large B-cell Lymphoma; Rituximab; Toripalimab
Keywords: DLBCL; CD20; Toripalimab; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combine with Rituximab (Experimental): Experimental: Toripalimab combine with Rituximab
  Induction period:
  Toripalimab 240mg administered intravenously (IV) on Day 1 of each 21-day cycle for 6 cycles.
  Rituximab 375mg/m² administered intravenously (IV) on Day 1 of each 21-day cycle for 6 cycles.
  Maintenance:
  Toripalimab 240mg administered intravenously (IV) and Rituximab 375mg/m² on Day 1 of each 56-day cycle for 6 cycles.
  Interventions: Drug: Toripalimab combine with Rituximab

INTERVENTIONS:
Drug: Toripalimab combine with Rituximab — Toripalimab is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2).
  Drug: Rituximab Rituximab is an antibody to CD20 molecules. One of the mechanisms of killing tumor cells is through antibody-dependent cell-mediated cytotoxicity (ADCC).
  Other Names: JS001 combine with rituxan

SUMMARY:
Exploring the efficacy and safety of Toripalimab with Rituximab for treatment of relapsed refractory CD20 positive diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Toripalimab is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2). Rituximab is an antibody to CD20 molecules. One of the mechanisms of killing tumor cells is through antibody-dependent cell-mediated cytotoxicity (ADCC). These two drugs may have a synergistic effect on anti-tumor. The purpose of this study is to determine whether Toripalimab with Rituximab is effective and safe for treatment of relapsed refractory CD20 positive diffuse large B-cell lymphoma. This is an exploratory small sample, phase II, single-center clinical trial, which is going to enroll 20 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. According to the WHO 2016 classification criteria, the CD20 positive diffuse large B-cell lymphoma (DLBCL) diagnosed by pathology should include the indicators of immunohistochemistry: CD10, BCL-2, MUM-1, BCL-6 and C-MYC;
3. Relapsed or refractory DLBCL.Patients younger than 65 years should relapse or progress after receiving at least second-line treatment, and patients 65 years of age and older could be intolerant to second-line treatment, and they who relapse or progress after receiving first-line treatment;
4. There is at least one measurable lesion, defined as measurable dual-diameter, intra-lymph node lesion, short diameter> 1.5cm, extra-lymph node lesion short diameter> 1.0cm;
5. Recurrence confirmed by pathological biopsy and CD20 positive;
6. ECOG score 0-2 points;
7. No autoimmune diseases;
8. Blood routine examination meets the following criteria:

   1. Neutrophil count ≥ 1.5 x 109 / L,;
   2. Platelet ≥ 75 x 109 / L,;
   3. Hemoglobin ≥ 10.0 g / dL;
9. The main organ function meets the following criteria:

   1. Aspartate aminotransferase and alanine aminotransferase ≤ 2.0 times the upper limit of normal value;
   2. Bilirubin ≤ 2.0 mg / dL;
   3. Creatinine clearance rate ≥ 60 mL / min;
10. Patients must agree to take effective contraceptive measures during the study according to the investigator's request;
11. Understand and voluntarily sign written informed consent.

Exclusion Criteria:

1. Diagnosed as transformed diffuse large B-cell lymphoma;
2. Diagnosed as double-hit diffuse large B-cell lymphoma (DHL);
3. Diagnosed as primary or secondary central nervous system lymphoma;
4. HBV DNA positive or HCV RNA positive patients;
5. Left ventricular ejection fraction <50%;
6. Patients with history of autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, Sjogren's syndrome, ankylosing spondylitis
7. Patients are using or have been used immunosuppressive drugs
8. Patients with ≥2 grade peripheral neuropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 24 months
  From the beginning of treatment, adopt Lugano 2014 evaluation standard, imaging examinations are performed every 2 cycles to assess changes in disease until progression or death
Progression Free Survival(PFS) | up to 24 months
  From the date into this study to disease progression or death

SECONDARY OUTCOMES:
To assessment of the safety events | up to 24 months
  Number of subjects experiencing different-grade toxicity
Assessment of the correlation between tumor cell PD-L1 expression intensity and efficacy | up to 24 months
  Subjects will be according to the Lugano 2014 criteria assessed with computed tomograph(CT) at screening,after completion of treantment therapy and during the post-treatment follow-up period.Baseline biopsies for immunologic analyses will be obtained from patients. Secondary histologic outcome include percent PD-L1 positive tumor cells by immunohistochemistry.

OTHER OUTCOMES:
Analysis of the correlation between the ammount of T cells and NK cells around tumor cells | up to 24 months
  Baseline and post-treatment biopsies for immunologic analyses will be obtained from patients.Histologic outcomes include percent and density PD-L1 positive tumor cells, percent and density CD56 postive NK cells, percent and density CD3 positive T cells by immunohistochemistry.
Change in immune microenviroment at the time of initial diagnosis and relapse | up to 24 months
  Immune mincroenviroment to be assessed by analyzing changes in the immune infiltrate in biopsy specimens obtained at initial diagnosis and relapse. Histologic outcome include percent and density PD-L1 positive tumor cells and CD3,CD4,CD8,CD56,CD58,PD-1,β2-MG,CIITA,HLA-DR/DP/DQ positive cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China